CLINICAL TRIAL: NCT01957514
Title: Intensive Trial of OMics in Cancer (ITOMIC) - Intensive Longitudinal Monitoring in Subjects With Triple-Negative Breast Cancer
Brief Title: Collecting, Analyzing, and Storing Samples From Patients With Metastatic, Triple Negative Breast Cancer Receiving Anti-cancer Therapy
Acronym: ITOMIC
Status: Terminated | Type: Observational
Why Stopped: Terminated due to loss of funding.
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 8132; NCI-2013-01654 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ITOMIC-001; UW13022; 8132 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1013004 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Stage IV Breast Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, buccal mucosa, saliva, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (sample collection): Patients undergo collection of tissue biopsy, blood, buccal swab, saliva, and urine at baseline.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo tissue biopsy, blood, buccal mucosa, saliva, and urine collection
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot research trial studies collecting, analyzing, and storing samples from patients with triple negative breast cancer (breast cancer cells that do not have estrogen receptors, progesterone receptors, or large amounts of human epidermal growth factor receptor 2 protein) that has spread to other places in the body receiving anti-cancer therapy. Studying samples of tissue, blood, buccal swab, saliva, and urine in the laboratory from patients receiving anti-cancer therapy may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety and feasibility of collecting, analyzing and storing clinically annotated panomic and other data from serially monitored subjects with metastatic triple negative breast cancer (TNBC) who receive care from up to ten oncology practices across the United States.

SECONDARY OBJECTIVES:

I. To determine whether molecular changes associated with resistance to treatment can be identified.

II. To understand subject perceptions regarding panomic data and its application to cancer treatment.

III. To apply other technologies to the characterization of subject tumors as they become available.

OUTLINE:

Patients undergo collection of tissue biopsy, blood, buccal mucosa, saliva, and urine at baseline. Additional biopsies may be performed prior to treatment change.

After completion of biopsy, patients are followed up at 1 day and 7 days. Patients will be followed indefinitely or for as long as they agree to be in the study, depending on the availability of resources.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have metastatic TNBC
* Disease suitable for analysis from either (a) or (b) below:

  * (a) Research biopsy

    * Tumor tissue, which can include bone disease, as determined by physical exam or imaging (as assessed by a trained specialist in radiology)
    * Must be collected before the subject receives treatment with a drug they have not received previously
  * (b) Standard of care biopsy

    * Tumor tissue available from a previous biopsy as standard of care (to be determined by the principal investigator [PI] or his designee)
    * Must have been collected before subject receives treatment with a drug they have not received previously
    * May begin treatment either after enrollment or within several weeks prior to enrollment
* Subjects must be medically fit and willing to undergo repeated tissue biopsies or surgical procedures to get tumor tissue
* Procedure-specific signed informed consent prior to initiation of any study-related procedures
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (or a Karnofsky performance status of >= 50%)
* Agree to allow their de-identified clinical and laboratory data to be posted to publicly available databases such as database of Genotypes and Phenotypes (dbGaP)

Exclusion Criteria:

* Bevacizumab treatment within 4 weeks prior to biopsy
* Anticoagulation therapy, unless reversed at the time of biopsy
* The enrolling study oncologist has decided that the subject is not fit enough to undergo repeated tissue biopsies
* Presence of a condition or abnormality that in the opinion of the enrolling investigator would compromise the safety of the subject or the quality of the data
* Significant bleeding disorder
* Known brain metastases that have not or will not be treated
* Subjects with a life expectancy of less than 6 months
* Prisoners
* Inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic TNBC treated at Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events resulting from performing multiple biopsies measured by the presence of biopsy-related complications, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Within 1 week of biopsy
  The frequency of adverse events associated with multiple repeated study-related biopsies (or leukapheresis runs) will be determined using simple statistics.
Infrastructure for acquiring, storing, retrieving and analyzing panomic data from clinical tumor specimens in a clinically relevant timeframe from participating sites | Up to 2 years
  Findings of potential clinical significance will be included in the reports provided to subjects and oncologists. Similarly, as new information becomes available, information of significance to understanding a subject's tumor or germline genomes may become apparent.

SECONDARY OUTCOMES:
Change in subject perceptions regarding panomic data and its application to cancer treatment assessed by Intensive Trial of OMics in Cancer baseline and follow up questionnaires | Baseline to 2 years
  Subject perceptions regarding the value of panomic testing in predicting the optimal treatment for subjects with cancer and for predicting the risk for developing other inherited diseases will be collected.
Develop process improvements | Up to 2 years
  The yield of successfully performing various types of analyses from clinically indicated- and study-related biopsies and leukapheresis specimens as well as the time frame necessary for returning reports will be monitored.
Development and improvement of infrastructure for storing and working with data from subject biopsies | Up to 2 years
  Data from subjects will be used to test the infrastructure being developing and identify areas that need to be improved.
Methods required to analyze and integrate data across subjects and with data from the public domain | Up to 2 years
  Methods and software that can facilitate comparing data from subjects with that deposited in the public domain will be developed.
Molecular changes associated with treatment response or resistance | Up to 2 years
  A number of statistical approaches will be used. Will be evaluated by comparing biopsies taken from the same subject pre- and post- anti-cancer treatment, and relating these changes to each subject's outcome.
Number or frequencies of biopsies or leukapheresis runs | Up to 2 years
  Safety and feasibility data will be analyzed and the frequency, nature, and severity of adverse events will be summarized.
Removal of any unnecessary biopsies or generation of redundant data | Up to 2 years
  Data across biopsies taken from the same individual at the same time point will be compared to assess the need for multiple biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Duan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington